CLINICAL TRIAL: NCT05670535
Title: Vaginal Infections and Sexual Dysfunction in Women With Primary Sjögren's Syndrome
Brief Title: Sjögren and Gynecologic Considerations
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Esin Merve Erol Koç, Medical Doctor, Obstetrician and Gynecologist, Principal Investigator, Ankara City Hospital Bilkent
Other Study IDs: E1-20-1290
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Primary Sjögren Syndrome; Vaginitis Candida; Vaginitis; Sexual Dysfunction
Keywords: Acute vaginitis; Dyspareunia; Gynecological complaints; Sexual dysfunction; Sjögren's Syndrome; Vaginal candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Vaginitis; Sexual Dysfunction, Physiological; Dyspareunia; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pSS group (Study group): * Women with the diagnosis of pSS for at least 3 years.
  * At reproductive age (without menopause).
  * Receiving only hydroxychloroquine sulfate treatment.
  * Presence of the symptoms of vaginitis.
  Interventions: Other: Visual analogue scale (VAS) for dyspareunia; Other: Visual analogue scale (VAS) for vaginal dryness; Other: The European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ESSDAI); Other: The European League Against Rheumatism Sjögren's Syndrome Patient Reported Index (ESSPRI)
- Women without pSS (Control group): * Women without any known disease.
  * At reproductive age (without menopause).
  * Presence of the symptoms of vaginitis.
  Interventions: Other: Visual analogue scale (VAS) for dyspareunia; Other: Visual analogue scale (VAS) for vaginal dryness; Other: The European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ESSDAI); Other: The European League Against Rheumatism Sjögren's Syndrome Patient Reported Index (ESSPRI)

INTERVENTIONS:
Other: Visual analogue scale (VAS) for dyspareunia — Dyspareunia scores between 0 to 10 points
Other: Visual analogue scale (VAS) for vaginal dryness — Vaginal dryness scores between 0 to 10 points
Other: The European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ESSDAI) — Sjögren's Syndrome Disease Activity Index scores between 0 to 3 points
Other: The European League Against Rheumatism Sjögren's Syndrome Patient Reported Index (ESSPRI) — Sjögren's Syndrome Patient Reported Index scores between 0 to 10 points

SUMMARY:
Sjögren's syndrome is an autoimmune disorder characterized by glandular and extra-glandular manifestations. It is called primary Sjögren's syndrome (pSS) in absence of another connective tissue disease. The hallmark symptoms of pSS are dry eyes and dry mouth due to the decreased lacrimal and salivary gland functions. However, other tissue and organs may also be involved which precede such as xerotrachea in upper airway, atrophic gastritis and pancreatitis in gastrointestinal tract, and dryness in vaginal mucosa.

Regarding to the genital involvement in pSS, vaginal dryness and resultant vaginal discomfort, and pain are reported as the common complaints. The transudate released by vaginal mucosa is the main resource of vaginal secretions.The human microbiome was reported to have a potential impact in etiopathogenesis of certain autoimmune disorders. The previous research revealed significant alterations in the gut, eye, and oral flora of the pSS patients. The disturbed oral flora due to immunodeficiency and reduced salivary flow was also reported to make the SS patients to prone to bacterial infections and recurrent oral candidiasis. Vaginitis has been defined as a spectrum of symptoms suggesting vulvovaginal discomfort such as itching, burning, irritation, and abnormal discharge. Even the vaginitis is an evidence of disturbance in vaginal flora, previous prospective research on vaginal microbiome of pSS patients either excluded the cases with vaginitis or not mentioned from the presence of vaginitis in women with pSS. To the best of our knowledge, there has not been any study yet to define the characteristics of vaginal flora through the presence of clinical signs and symptoms in women with pSS. To gain more insight into the clinical context of the gynecologic complaints, sexual dysfunction, and presence of vaginitis in pSS, the current study aims to identify the associations between these issues and pSS related disease parameters.

DETAILED DESCRIPTION:
Sjögren's syndrome is an autoimmune disorder characterized by glandular and extra-glandular manifestations. In the absence of another connective tissue disease, it is called primary Sjögren's syndrome (pSS). The hallmark symptoms of pSS are dry eyes and dry mouth due to the decreased lacrimal and salivary gland functions. However, other tissue and organs may also be affected including the vaginal mucosa. Regarding to the genital involvement in pSS, vaginal dryness and resultant vaginal discomfort, and pain are reported as the common complaints. The transudate released by vaginal mucosa is the main resource of vaginal secretions.The human microbiome was reported to have a potential impact in etiopathogenesis of certain autoimmune disorders. The previous research revealed significant alterations in the gut, eye, and oral flora of the pSS patients. The disturbed oral flora due to immunodeficiency and reduced salivary flow was also reported to make the SS patients to prone to bacterial infections and recurrent oral candidiasis. Vaginitis has been defined as a spectrum of symptoms suggesting vulvovaginal discomfort such as itching, burning, irritation, and abnormal discharge. Even the vaginitis is an evidence of disturbance in vaginal flora, previous prospective research on vaginal microbiome of pSS patients either excluded the cases with vaginitis or not mentioned from the presence of vaginitis in women with pSS. To the best of our knowledge, there has not been any study yet to define the characteristics of vaginal flora through the presence of clinical signs and symptoms in women with pSS. To gain more insight into the clinical context of the gynecologic complaints, sexual dysfunction, and presence of vaginitis in pSS, the current study aims to identify the associations between these issues and pSS related disease parameters. In this prospective cohort study, we planned to include sexually active 118 women at reproductive age who had the symptoms of itching, burning, irritation, and abnormal discharge. Women with pSS (study group, n=49) will be compared with women who had not any other disease or complaint rather than vaginal discharge (control group, n=69). Besides the physical examination and gynecological evaluation including sterile speculum examination enabling swab sampling for vaginal discharge and PAP smear; the Visual analogue scales (VAS) for dyspareunia, and vaginal dryness and The European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ESSDAI), and Sjögren's Syndrome Patient Reported Index (ESSPRI) Sjögren's syndrome disease activity will be also performed. Correlation and regression analyses will be also performed for pSS related parameters.

ELIGIBILITY:
Inclusion Criteria:

* All participants are recruited from women who consecutively applied to outpatient clinic.
* Normally menstruating women at reproductive age (without menopause) for all participants.
* Regular sexual activity with single sexual partner for all participants.
* Receiving only hydroxychloroquine sulfate treatment for women with pSS.
* Presence of the symptoms of vaginitis for all participants.
* Without any known disease including autoimmune disorders for women in control group.

Exclusion Criteria:

* Women with the pelvic anatomical structural abnormalities
* History of any type of cancer including gynecological cancers, chemotherapy, and/or radiotherapy,
* Endometriosis, chronic cervicitis, menopause, pregnancy, lactation, use of hormonal contraceptive medication, use of vaginal estrogen, pre-malign or malign cytology at Papanicolaou (PAP) smear, having intrauterine device,
* Smoking,
* Chronic diseases (diabetes mellitus, psychiatric disorders,
* Multiple sexual partners, sexually transmitted infections including gonorrhea, chlamydia, genital herpes, and/or mycoplasma, mixed vaginal infections,
* Urinary tract infection in last three months,
* Antibiotic medication at last one month,
* Administration of drugs which may lead vaginal dryness including antihistaminics, antidepressants, and anti-hypertensives,
* Treatment with glucocorticoids, biologic disease modifying anti-rheumatic drugs, or immune-suppressive agents at last three months
* Women who had sexual partners with any sexual dysfunction

Ages: 20 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: This study is designed as a prospective cohort study, to include sexually active 118 women at reproductive age who had the symptoms of itching, burning, irritation, and abnormal discharge. Women with pSS (study group, n=49) will be compared with women who had not any other disease or complaint rather than vaginal discharge (control group, n=69). All the participants will be recruited from sexually active women with single sexual partner.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Vaginal candidiasis | 20 minutes
  Culture of swab sampling from vaginal fluid at Sabouraud dextrose agar plates incubated in CO2 for evaluation of candida
Acute vaginitis | 10 minutes
  Laboratory assessment of vaginal swab sampling from vaginal fluid for bacterial vaginosis
Visual analogue scale for dyspareunia | 20 minutes
  The severity of symptoms scored between 0 (no symptoms) to 10 (worst symptoms) points.
Visual analogue scale for vaginal dryness | 20 minutes
  The severity of symptoms scored between 0 (no symptoms) to 10 (worst symptoms) points.
The European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ESSDAI) | 20 minutes
  The severity of clinical signs regarding Sjögren's Syndrome disease activity, scored between 0 (no symptoms) to 3 (worst symptoms) points.
The European League Against Rheumatism Sjögren's Syndrome Patient Reported Index (ESSPRI) | 20 minutes
  he severity of patient reported symptoms regarding Sjögren's Syndrome, scored between 0 (no symptoms) to 10 (worst symptoms) points.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The research data is not shared unless it is needed.

REFERENCES:
- [Result] Mariette X, Criswell LA. Primary Sjogren's Syndrome. N Engl J Med. 2018 Mar 8;378(10):931-939. doi: 10.1056/NEJMcp1702514. No abstract available. PMID 29514034
- [Result] Priori R, Minniti A, Derme M, Antonazzo B, Brancatisano F, Ghirini S, Valesini G, Framarino-dei-Malatesta M. Quality of Sexual Life in Women with Primary Sjogren Syndrome. J Rheumatol. 2015 Aug;42(8):1427-31. doi: 10.3899/jrheum.141475. Epub 2015 Jul 1. PMID 26136488
- [Result] Mulherin DM, Sheeran TP, Kumararatne DS, Speculand B, Luesley D, Situnayake RD. Sjogren's syndrome in women presenting with chronic dyspareunia. Br J Obstet Gynaecol. 1997 Sep;104(9):1019-23. doi: 10.1111/j.1471-0528.1997.tb12060.x. PMID 9307528
- [Result] Brito-Zeron P, Baldini C, Bootsma H, Bowman SJ, Jonsson R, Mariette X, Sivils K, Theander E, Tzioufas A, Ramos-Casals M. Sjogren syndrome. Nat Rev Dis Primers. 2016 Jul 7;2:16047. doi: 10.1038/nrdp.2016.47. PMID 27383445
- [Result] ACOG Committee on Practice Bulletins--Gynecology. ACOG Practice Bulletin. Clinical management guidelines for obstetrician-gynecologists, Number 72, May 2006: Vaginitis. Obstet Gynecol. 2006 May;107(5):1195-1206. doi: 10.1097/00006250-200605000-00049. PMID 16648432